CLINICAL TRIAL: NCT04033796
Title: Vitamin D Supplementation in the Armed Forces (D_SAF) PILOT STUDY
Brief Title: Vitamin D Supplementation D_SAF Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: Institute of Naval Medicine (Unknown); CTRM Lympstone (Unknown); Navy Command Headquarters (Unknown)
Responsible Party: Principal Investigator, Susan Lanham-New, Professor, University of Surrey
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: D_SAF Pilot study
Record Dates: First submitted 2019-07-23; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 25,000 IU (Active Comparator)
  Interventions: Dietary Supplement: 25,000 IU
- 50,000 IU (Active Comparator)
  Interventions: Dietary Supplement: 50,000 IU
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 25,000 IU — Vitamin-D3 supplementation providing 25,000 IU administered orally every two months (equivalent to ~400 IU/d);
  Arms: 25,000 IU
Dietary Supplement: 50,000 IU — Vitamin-D3 supplementation providing 50,000 IU administered orally every two months (equivalent to ~800 IU/d);
  Arms: 50,000 IU
Dietary Supplement: Placebo — A placebo (administered orally every two months) supplementation control group.
  Arms: Placebo

SUMMARY:
This study is a randomised control trial (RCT) pilot study to determine the appropriate vitamin D dose for the main study. The pilot study includes three matched groups, which will form two vitamin D supplementation groups (at 25,000 IU and 50,000 IU every two months), and a third placebo supplementation group. The aim was to develop an appropriate supplementation regimen that was compatible with recruit training and maintained serum vitamin D (25OHD) status above 50 nmol/l during recruit training.

DETAILED DESCRIPTION:
Study Overview:

Aim: The dose-response to vitamin D3 supplementation in Royal Marine recruits undertaking military training. Part-A of this research project will provide a pilot study for the main study. Volunteer recruits will initially complete a healthy history, smoking habit and alcohol consumption questionnaire. Height, body mass (from which BMI will be calculated), and calf girth/skinfold will be measured. A 20 ml blood sample will be drawn in two parts: a 15 ml blood sample (gold top serum vacutainers) for determination of vitamin D status, calcium and albumin concentrations, PTH levels, serum collagen type I cross-linked C-telopeptide (CTx), carboxy-terminal propeptide of type I collagen (P1NP), ferritin (Fe) and antibody responses against S. aureus or other antigens; and a 5 ml blood sample (white top EDTA plasma vacutainers) will be drawn for determination of plasma cytokine levels. At one sample point only, DNA will be extracted from the cell pellet acquired following centrifuging of the whole blood to separate the plasma. This DNA will be analysed for the specific single nucleotide polymorphisms (SNPs) that have been shown to be associated with vitamin D metabolism. Permission will also be sought to collate the outcome of the week-1 and week-9 Royal Marine Fitness Assessment (RMFA). The pilot study recruit cohort will be randomised into one of three groups: (i) a vitamin-D3 supplementation providing 25,000 IU administered orally every two months (equivalent to ~400 IU.d-1); (ii) a vitamin-D3 supplementation providing 50,000 IU administered orally every two months (equivalent to ~800 IU.d-1); and (iii) a placebo (administered orally every two months) supplementation control group. The vitamin D and placebo supplements will be manufactured by Pharmaterials Ltd., Unit B, 5 Boulton Road, Reading, RG2 0NH, UK. Both the active and placebo supplements will be presented as identical (size and appearance) tablets, indiscernible from each other for either the volunteer or the study team in situ at CTC. All three groups will receive one tablet at each time point. Recruits will be randomly assigned to a study group, but the three groups will be matched for age, height, body mass and aerobic fitness. Randomisation of supplement/placebo administration to study volunteers will be undertaken by Statisticians from the University of Surrey. Study team staff will monitor supplement taking and will further confirm supplement taking through exit interviews. Further 20 ml blood samples will be drawn every two months (i.e. at weeks 8, 16 and 32 of RM training), and the smoking habit and alcohol consumption questionnaire will be readministered. The Food Frequency Questionnaire (FFQ)25,26 will be administered in week- 6 of training; this will allow the recruits' habitual RM training diet to be established following the civilian to military transition. Permission will be sought to collate the outcome of the week-1 and week-9 Royal Marine Fitness Assessment (RMFA). Permission will also be sought to prospectively collate data from the Defence Medical Information Capability Programme (DMICP) system describing the prevalence of injury and illness in study volunteers.

ELIGIBILITY:
Inclusion Criteria:

* RM recruit troops commencing training during the winter and summer months,
* aged between 16 - 32 years at the Start of Training
* having successfully completed the physical and professional selection tests which comprise the Potential Royal Marine Course (PRMC)
* be deemed medically fit and healthy following medical screening at the AFCO and again at CTC if required

Exclusion Criteria:

* not participating in Recruit Syllabus (RS10) for RM recruit training
* deemed unsuitable by the IMO or the training team

Ages: 16 Years to 32 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 532 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-06-10 (Actual); Study Completion 2016-06-10 (Actual)

PRIMARY OUTCOMES:
The dose-response changes in 25-hydroxyvitamin D | 32 weeks
The incidence of injury/illness in recruits during training | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L Fallowfield, PhD, Principal Investigator — Institute of Naval Medicine; Susan A Lanham-New, Professor, Principal Investigator — University of Surrey
Locations (2):
- United Kingdom (2):
  - University of Surrey, Guildford, Surrey
  - Institute of Naval Medicine, Gosport

IPD SHARING:
Plan to Share IPD: No